CLINICAL TRIAL: NCT02641314
Title: Phase 2 Trial of Metronomic Treatment in Children and Adolescents With Recurrent or Progressive Neuroblastoma (NB)
Brief Title: Metronomic Treatment in Children and Adolescents With Recurrent or Progressive High Risk Neuroblastoma
Acronym: METRO-NB2012
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Marc Hömberg, Dr., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1495; 2011-004593-29 (EudraCT Number)
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Neuroblastoma
Keywords: Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Administration, Metronomic; Propranolol; Celecoxib; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metronomic therapy (Experimental): Treatment consists of eight alternating 28-day-cycles of propranolol, celecoxib, cyclophosphamide, vinblastine, etoposide (PCCVE) and of propranolol, celecoxib, cyclophosphamide, vinblastine (PCCV) followed by five cycles PCCV resulting in a total of 13 cycles (364 days of treatment)
  Interventions: Drug: metronomic therapy

INTERVENTIONS:
Drug: metronomic therapy — * Propranolol 0.5 mg/kgxd p.o. day 1,
    1. mg/kgxd p.o. day 2,
    2. mg/kgxd p.o. day 3-365 (maximum total daily dose: 120 mg) divided in 2 doses per day
  * Celecoxib 400 mg/m2xd p.o.; day 1-365 (maximum total daily dose: 800 mg) divided in 2 doses per day
  * Cyclophosphamide cycle 1, day1: loading dose: 500 mg/m2 intravenous 1-h-infusion, single dose day 2-365 25 mg/m2xd p.o (maximum total daily dose: 50 mg) as single daily dose
  * Vinblastine 3 mg/m2xd i.v. (maximum total daily dose: 6 mg) administered day 1 and 15 (every two weeks) as single daily dose
  * Etoposide 25 mg/m2xd p.o.; day 1-21 weeks 1-3, 9-11, 17-19, 25-27 (maximum total daily dose: 50 mg) as single daily dose
  Other Names: Dociton; Celebrex; Endoxan; Lastet; Vinblastinsulfat Teva

SUMMARY:
Neuroblastoma is the second most frequent cause for death from cancer in childhood. Already one year after diagnosis of recurrence from high risk neuroblastoma, 75% of the patients experience further progression.

Metronomic therapy is targeting not only the tumor cell, but also the tumor supplying vasculature and the interactions between Tumor and immune cells. The toxicity is expected to be low due to the low (but continuous) dosing of drugs.

The study investigates the tolerance and the efficacy of a new combination of five drugs consisting of propranolol (antiangiogenetic, anti-neuroblastic), Celecoxib (modulating immune response, ant-neuroblastic), cyclophosphamide (antiangiogenetic, anti-neuroblastic), etoposide (antiangiogenetic, anti-neuroblastic), and vinblastin (antiangiogenetic, anti-neuroblastic). Vinblastin is scheduled every 14 days intravenously, all other drugs are applied daily throughout 365 days (except etoposide for 4x3 weeks). The efficacies of each of the drugs have been demonstrated in vitro and in vivo in animal studies. All drugs have been used in children for other conditions. From those experiences low toxicities and a favorable Quality of life are expected.

DETAILED DESCRIPTION:
Neuroblastoma relapses during or after intensive therapy most likely result from the presence of primary or acquired drug resistance. Therefore, new therapeutic modalities for salvage therapies are urgently needed.

The historical Kaplan-Meier curves of 218 unselected high risk patients after the first recurrence (from CR) or after the first progression (from PR/SD) demonstrate a 1 year event free survival rate of 25.2 ± 2.9% and a 1 year overall survival rate of 42.7 ± 3.3%.

Today cancer is widely considered as a multicomponent disease. One novel strategy likely to target the complexity of tumor cells and tumor environment is metronomic scheduling of anticancer treatment or "metronomic treatment" (MT). Low doses of chemotherapeutic drugs are continuously administered to cancer patients. The higher frequency and lower dose targets distinct aspects of cancer's functionality. Effects on tumor-angiogenesis, anti-cancer immunity and tumor stroma have been shown. Additionally low-dose metronomic treatment is often combined with modern antiinflammatory or antiangiogenic drugs, which specifically interact e.g. in tumor growth or angiogenesis pathways.

The rationale of this trial is the efficacy of metronomic therapy in heavily pre-treated refractory neuroblastoma patients.This trial protocol proposes a metronomic schedule of low dose chemotherapy with cyclophosphamide, etoposide and vinblastine, in combination with propranolol, a non-selective blocker of β adrenergic receptors and celecoxib, a selective cyclooxygenase type 2 (COX-2) inhibitor.

Patients enrolled in this study may benefit for two reasons. In the palliative situation, metronomic treatment may result in disease stabilization (SD) and a significant improvement of the quality of life (QOL) of patients e.g. by the decrease of pain through the treatment. For this reason, QOL including pain module is assessed as a separate secondary objective/ outcome measure. In the case of tumor response (PR, CR), the patients may qualify for a subsequent treatment approach aiming at further disease stabilization or even a long-term benefit.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed recurrence or progression of high risk neuroblastoma which progressed despite previous treatment (irrespective of the number of previous relapses/progressions).
* Refractory and/or residual high-risk neuroblastoma with measurable or evaluable disease irrespective of preceding treatment (no Progression during the minimal interval as defined below)
* Age: ≥ 2 years and < 21 years
* Measurable or evaluable disease defined as

  * Presence of at least one measurable (recurrent or newly progressing) neuroblastoma lesion ≥ 10 mm by magnetic resonance imaging (MRI) or computed tomography (CT) or
  * Newly detected unambiguous scintigraphic (MIBG) avid bone and/or medullary lesions
  * presence of unambiguous bone marrow metastasis
* Minimal interval between start of trial medication and preceding anti-cancer treatment is 4 weeks after chemotherapy, 6 weeks after radiotherapy, and 12 weeks after myeloablative therapy
* Life expectancy > 3 months
* Good to moderate general condition (performance scale ≥60)
* No serious infection
* Spontaneous recovering blood counts:

  * White blood cell count ≥ 1000/µL
  * Neutrophil count ≥ 500/µL
  * Platelet count ≥ 25 000/µL (unsupported)
* Written informed consent of parents or legal guardian and/ or patient according to age and status of psycho-intellectual development.

Exclusion Criteria:

* Minimal residual disease status (only) without unambiguous measurable or evaluable disease
* Patients unable to swallow trial medication
* Any concomitant anti-cancer treatment (e.g. other cytostatic drugs, "small molecules", antibodies, radiotherapy, surgery of tumor or metastases)
* Treatment with medication that interact with study medication that cannot be discontinued at least one week prior to the start of trial medication and for the duration of the trial
* Intake of antihypertensive drugs, e.g. calcium channel blockers
* Established hypersensitivity to the active or one of the other constituents of the trial medication
* Severe medical or psychosocial conditions preventing trial participate and/or any of the following

  * Peripheral neuropathy or constipation CTCAE grade 3 or 4
  * Cardiac arrhythmias (sinus bradycardia for age, sinus arrhythmia as 2.-3. grade atrioventricular block)
  * Pre-existing recurrent symptomatic bronchial asthma
  * Diabetes mellitus (propranolol covers symptoms of hypoglycemia)
  * Conditions with low blood pressure below age-dependent normal ranges
  * History of gastrointestinal ulcer or perforation
  * Known active hepatitis B virus (HBV), hepatitis C (HBC) virus or human immunodeficiency virus (HIV) infection
* Concomitant participation in other clinical trials with investigational drugs or with competing interventions
* Pregnancy, lactation
* Sexually active patients not willing to use highly effective contraception

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
non-inferiority of EFS compared to historical control group | up to 12 months
  The primary trial objective is to demonstrate the non-inferiority of event free survival (EFS) in comparison to a historical control group. Event free survival (EFS) defined as time from start of treatment up to Progression (emerged from residual tumor, PD) or recurrence (developing from CR achieved by metronomic treatment), permanent discontinuation of treatment for unacceptable toxicity, secondary malignant neoplasm or death of any reason.

SECONDARY OUTCOMES:
disease control rate at 6 months | 6 months after start of treatment
  Disease control rate at 6 months of metronomic treatment defined as number of patients achieving overall complete response (CR), partial response (PR) or stable disease (SD) related to all treated patients.
Overall survival | up to 12 months
  Overall survival defined as time from start of treatment until death of any reason or date of last information
hospitalization days | up to 395 days
  Any patient stay in hospital that includes at least one night from day 1 of metronomic treatment until 30 days after the end of treatment. Overall treatment time is 12 months.
number of transfusion days | up to 365 days
  The number of days with transfusion of platelets or packed red blood cells. Overall treatment time is 12 months.
drop-out rate | up to 12 months
  The number and rate of patients stopping metronomic treatment during treatment period due to patients and/or parents wish. Overall treatment time is 12 months.
disease control rate at 12 months | 12 months after start of treatment
  Disease control rate at 12 months of metronomic treatment defined as number of patients achieving overall complete response (CR), partial response (PR) or stable disease (SD) related to all treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Hoemberg, Dr., Principal Investigator — University of Cologne
Locations (8):
- Germany (8):
  - Children's University Hospital, Bonn
  - Marc Hoemberg, Cologne
  - Children's University Hospital, Essen
  - Children's University Hospital, Frankfurt
  - Children's University Hospital, Freiburg im Breisgau
  - Children's Hospital, Medizinische Hochschule, Hanover
  - Children's University Hospital, Leipzig
  - Dr. von Haunersches Kinderspital, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simon T, Berthold F, Borkhardt A, Kremens B, De Carolis B, Hero B. Treatment and outcomes of patients with relapsed, high-risk neuroblastoma: results of German trials. Pediatr Blood Cancer. 2011 Apr;56(4):578-83. doi: 10.1002/pbc.22693. Epub 2010 Dec 9. PMID 21298742
- [Background] Klement G, Baruchel S, Rak J, Man S, Clark K, Hicklin DJ, Bohlen P, Kerbel RS. Continuous low-dose therapy with vinblastine and VEGF receptor-2 antibody induces sustained tumor regression without overt toxicity. J Clin Invest. 2000 Apr;105(8):R15-24. doi: 10.1172/JCI8829. PMID 10772661
- [Background] Ghiringhelli F, Menard C, Puig PE, Ladoire S, Roux S, Martin F, Solary E, Le Cesne A, Zitvogel L, Chauffert B. Metronomic cyclophosphamide regimen selectively depletes CD4+CD25+ regulatory T cells and restores T and NK effector functions in end stage cancer patients. Cancer Immunol Immunother. 2007 May;56(5):641-8. doi: 10.1007/s00262-006-0225-8. Epub 2006 Sep 8. PMID 16960692
- [Background] Wang YC, He F, Feng F, Liu XW, Dong GY, Qin HY, Hu XB, Zheng MH, Liang L, Feng L, Liang YM, Han H. Notch signaling determines the M1 versus M2 polarization of macrophages in antitumor immune responses. Cancer Res. 2010 Jun 15;70(12):4840-9. doi: 10.1158/0008-5472.CAN-10-0269. Epub 2010 May 25. PMID 20501839
- [Background] Ponthan F, Wickstrom M, Gleissman H, Fuskevag OM, Segerstrom L, Sveinbjornsson B, Redfern CP, Eksborg S, Kogner P, Johnsen JI. Celecoxib prevents neuroblastoma tumor development and potentiates the effect of chemotherapeutic drugs in vitro and in vivo. Clin Cancer Res. 2007 Feb 1;13(3):1036-44. doi: 10.1158/1078-0432.CCR-06-1908. PMID 17289900
- [Background] Nakanishi Y, Nakatsuji M, Seno H, Ishizu S, Akitake-Kawano R, Kanda K, Ueo T, Komekado H, Kawada M, Minami M, Chiba T. COX-2 inhibition alters the phenotype of tumor-associated macrophages from M2 to M1 in ApcMin/+ mouse polyps. Carcinogenesis. 2011 Sep;32(9):1333-9. doi: 10.1093/carcin/bgr128. Epub 2011 Jul 5. PMID 21730361
- [Background] Asgharzadeh S, Salo JA, Ji L, Oberthuer A, Fischer M, Berthold F, Hadjidaniel M, Liu CW, Metelitsa LS, Pique-Regi R, Wakamatsu P, Villablanca JG, Kreissman SG, Matthay KK, Shimada H, London WB, Sposto R, Seeger RC. Clinical significance of tumor-associated inflammatory cells in metastatic neuroblastoma. J Clin Oncol. 2012 Oct 1;30(28):3525-32. doi: 10.1200/JCO.2011.40.9169. Epub 2012 Aug 27. PMID 22927533
- [Background] Pasquier E, Street J, Pouchy C, Carre M, Gifford AJ, Murray J, Norris MD, Trahair T, Andre N, Kavallaris M. beta-blockers increase response to chemotherapy via direct antitumour and anti-angiogenic mechanisms in neuroblastoma. Br J Cancer. 2013 Jun 25;108(12):2485-94. doi: 10.1038/bjc.2013.205. Epub 2013 May 21. PMID 23695022
- [Background] Andre N, Carre M, Pasquier E. Metronomics: towards personalized chemotherapy? Nat Rev Clin Oncol. 2014 Jul;11(7):413-31. doi: 10.1038/nrclinonc.2014.89. Epub 2014 Jun 10. PMID 24913374
- [Background] Berthold F, Homberg M, Proleskovskaya I, Mazanek P, Belogurova M, Ernst A, Sterba J. Metronomic therapy has low toxicity and is as effective as current standard treatment for recurrent high-risk neuroblastoma. Pediatr Hematol Oncol. 2017 Aug;34(5):308-319. doi: 10.1080/08880018.2017.1373314. Epub 2017 Nov 17. PMID 29148865